CLINICAL TRIAL: NCT03130595
Title: West Sweden Parkinson Objective Measurement Registry Study - an Observational Cohort Study of the Prevalence and Development of Motor Symptoms Assessed With Automated Accelerometry in People With Parkinson's Disease in West Sweden
Brief Title: West Sweden Parkinson Objective Measurement Registry Study
Acronym: WestPORTS
Status: Active, not recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Filip Bergquist, Associate Professor, Sahlgrenska University Hospital
Other Study IDs: WestPORTS; PARKreg (Registry Identifier: Svenska Parkinsonregistret)
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Parkinsonism; Parkinsonian Disorders
Keywords: accelerometry; Parkinson Kinetigraph
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PD outpatients in West Sweden: Cross-sectional random sample of patients with PD that have visited outpatient clinics in West Sweden in the last 6+6 months

SUMMARY:
WestPORTS will recruit a randomly selected population consisting of 25% of all individuals with Parkinson's disease (ICD G209) that have visited any of the seven major outpatient neurology or geriatrics clinics in West Sweden (population 1.7M) during a predefined 12 month period between Sept 2016 and April 2018.

Baseline clinical and demographic data will be collected along with a 6 x 24h accelerometry recording using the Parkinson Kinetigraph (Global Kinetics). Repeated data collections will be made with regular intervals of up to 2 years as long as subjects are alive and willing.

DETAILED DESCRIPTION:
The following data will be collected at baseline:

Date of birth Handedness Family history of Parkinson's disease Time of first motor symptom onset Laterality of symptom onset Time of diagnosis Time of first pharmacological intervention (if applicable) First antiparkinsonian drug

The following data will be collected at every visit/update Current living conditions Current non motor complications Current medications Hoehn and Yahr staging Clinical Impression of Severity Index in Parkinson's disease (CISI-PD)

Patient self assessments: PDQ8, NMS-Questionnaire, EQ5D-5L, Patient Reported Outcome in Parkinson's Disease (PRO-PD)

Parkinson Kinetigraph (PKG) accelerometry based recording of spontaneous movement patterns over a 6x24h period. The following indices will be extracted: median bradykinesia score (BKS), median dyskinesia score (DKS), Fluctuation Dyskinesia Score (FDS), Percent daytime with Immobility (PTI%), Percent daytime with tremor (PTT%).

The primary analysis will be descriptive and include demographic composition of the population, clinical characteristics and objective measurement data. In addition to indices a standardized qualitative assessment of PKG recordings will be made to identify motor fluctuations. Correlations between clinical ratings, patient reported outcomes, disease duration, age, medication and objective measurement indices will be studied

In the prospective phase of the study the development of objective movement recordings will be studied along with the development of clinical ratings and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Medical record with a G209 (Parkinson's disease) diagnosis
* A visit to one of the participating outpatient clinics in West Sweden within the last 6 months
* Informed consent

Exclusion Criteria:

* Diagnosis revised before visit.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25% of the population described by the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Objective measurement of spontaneous movement patterns | 144 hours
  Parkinson Kinetigraph

CONTACTS AND LOCATIONS:
Overall Officials: Filip Bergquist, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Clinical registry data will be immediately available as part of the national Parkinson Registry. Study specific data from objective measurements will be made available within the registry one year after final subject has been recruited. Access to data requires ethical permission and permission from the registry scientific committee SWEPAR.
Supporting Information: Study Protocol
Time Frame: See plan description
Access Criteria: Access to data requires ethical permission and permission from the registry scientific committee SWEPAR.
URL: http://www.neuroreg.se/